CLINICAL TRIAL: NCT03060434
Title: Prospective Controlled Crossover Study of the Role of Pentoxifylline in the Management of Lumbar Radiculopathy
Brief Title: Pentoxifylline and Lumbar Radiculopathy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, Dr Joseph Maarrawi, Associate Professor : Researcher - Pain Specialist - Neurosurgeon, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pento-LR
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Radiculopathy; Lumbar Disc Herniation; Lumbar Disc Disease
Keywords: pentoxifylline; Disc hernia; sciatica; lumbar radiculopathy
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Displacement; Intervertebral disc disease; Sciatica | interventions — Pentoxifylline; Ibuprofen; Acetaminophen; Pregabalin

STUDY DESIGN:
Intervention Model Description: Each patient will receive for 1 month: Ibuprofen 600 mg bid; Paracetamol 1g tid if needed; pregabalin 75 mg bid pentoxifylline 400 mg bid will be added for either the first or second 15 days (randomization)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor and the investigator are unaware of the sequence of the 15 days treatment with pentoxifylline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Ibuprofen
  Interventions: Drug: Ibuprofen
- Pentoxifylline (Experimental): Pentoxifylline oral tablets
  Interventions: Drug: Pentoxifylline Oral Tablet

INTERVENTIONS:
Drug: Pentoxifylline Oral Tablet — patient will receive for 15 days: Ibuprofen 600 mg bid; pregabalin 75 mg bid; paracetamol 1 g tid; pentoxifylline 400 mg bid
  Other Names: Ibuprofen; Paracetamol; pregabalin
  Arms: Pentoxifylline
Drug: Ibuprofen — patient will receive for 15 days: Ibuprofen 600 mg bid; pregabalin 75 mg bid; paracetamol 1 g tid
  Other Names: Paracetamol; pregabalin
  Arms: Control

SUMMARY:
The objective of this prospective controlled crossover study is to evaluate the efficacy and safety of pentoxifylline per os (800 mg daily) in the management of lumbar radiculopathy

DETAILED DESCRIPTION:
Patients with lumbar radiculopathy, are recruited from senior author clinic. After verification of inclusion and exclusion criteria, patients consenting to enter the study are given 2 sequences (order randomly assigned) of treatment: Ibuprofen 600 mg bid, with paracetamol 1000 mg tid, pregabalin 75 mg bid for 15 days with pentoxifylline and 15 days without it. Basic clinical and demographical data are noted. Lumbar MRI results are also noted. Clinical evaluation of the patient is performed and included: clinical examination (including motor exam of lower limbs); pain is assessed according to Numerical rating Scale (NRS), and relative percentage of global improvement.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lumbar radiculopathy
* Disc hernia confirming the diagnosis with radio-clinical concordance

Exclusion Criteria:

* Radicular deficit needing surgery
* Cauda equine syndrome
* Absence of radio-clinical concordance on MRI
* Contraindication for anti-inflammatory (Hypertension, renal insufficiency, gastric ulcer …)
* Previous intolerance to pentoxifylline, and/or to pregabalin and/or paracetamol
* Pregnancy
* Follow-up not possible
* Hepatic dysfunction
* History of drug abuse
* Current use of tramadol, codeine and/or morphine and its derivative
* Antidepressant use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | At day 15 (and Day 30)
  Pain assessment by NRS

SECONDARY OUTCOMES:
Patient global impression of improvement scale | day 15 and 30
  pain improvement scale from 1 to 7
Side effects | Day 15 and 30
  Reporting side effects by patient

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Maarrawi, MD, PhD, Principal Investigator — Hotel Dieu de France Hospital - Beirut, Lebanon, 16 6830
Locations (1):
- Hotel Dieu de France Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No